CLINICAL TRIAL: NCT06996678
Title: Investigation of the Effect of Virtual Reality on Cognitive Skills in Children With Attention Deficit Hyperactivity Disorders
Brief Title: Effect of Virtual Reality on Cognitive Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Leyla Kaya Ozturk, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HÜ-OT-LKO-04
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Virtual Reality
Keywords: Attention deficit and hyperactivity disorder; cognitive functions; motor skills; Virtual Reality
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: Two groups with an intervention group and a control group
Who Masked: Outcomes Assessor
Masking Description: The therapist who conducted the assessment tests was unaware of the participants' group assignments (interventon or control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin (intervention group) (Active Comparator): The intervention group will receive both occupational therapy and virtual reality.a) Occupational Therapy: The basis of OT intervention consisted of activities requiring increased attention, behavioral regulation, organizational skills, multiple cognitive skills, and motor skills.
  Virtual Reality: The virtual reality system consists of a camera, television, Eye Toy Play CD and Play Station 2. It is based on the principle of capturing movements represented in a virtual environment (Gatica and Méndez, 2014). In the Eye Toy system, individuals can see themselves on the screen through the camera. In this way, the person constantly interacts with the movements and challenges brought by video games. We can simply call the Eye Toy system a webcam with a motion sensor and microphone. The individual's position in the game is determined on the screen and can perceive the person according to the movements he/she exhibits.
  Interventions: Behavioral: virtual Reality; Behavioral: occupational therapy
- Plasebo (control group) (Active Comparator): The control group will receive occupational therapy. Occupational Therapy: The basis of OT intervention consisted of activities requiring increased attention, behavioral regulation, organizational skills, multiple cognitive skills, and motor skills.
  Interventions: Behavioral: occupational therapy

INTERVENTIONS:
Behavioral: virtual Reality — Virtual Reality: The virtual reality system consists of a camera, television, Eye Toy Play CD and Play Station 2. It is based on the principle of capturing movements represented in a virtual environment (Gatica and Méndez, 2014). In the Eye Toy system, individuals can see themselves on the screen through the camera. In this way, the person constantly interacts with the movements and challenges brought by video games. We can simply call the Eye Toy system a webcam with a motion sensor and microphone. The individual's position in the game is determined on the screen and can perceive the person according to the movements he/she exhibits. The main skills required by the games are; target-based movement, visuomotor skills, praxis and thinking process skills.
  Arms: Aspirin (intervention group)
Behavioral: occupational therapy — Occupational Therapy: The basis of OT intervention consisted of activities requiring increased attention, behavioral regulation, organizational skills, multiple cognitive skills, and motor skills

SUMMARY:
The aim of this study is to investigate the effects of virtual reality (VR) intervention on cognitive skills in children with attention deficit hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
The study was designed as a randomized controlled trial. A simple randomization method will be used to randomly assign individuals to two groups (intervention and control groups). A simple randomization method will be used where the intervention and control group papers are selected from a sealed envelope. Following the initial assessment of each participant, one of the papers labeled "intervention" or "control" will be randomly selected. This decision will determine whether the individual will be assigned to the intervention or control group. The study will be conducted at Hacettepe University. The intervention group will receive occupational therapy (OT) for 30 minutes once a week for 8 weeks and will play a virtual reality (VR) game with the Sony PlayStation 2 Eye Toy system for 20 minutes. Both the intervention and control groups will receive occupational therapy for only 30 minutes once a week for 8 weeks. The Dynamic Occupational Therapy Cognitive Assessment (DOTCA-Ch) will be administered before and after the intervention to assess children's cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 7-12, having diagnosed with ADHD by a child psychiatrist in accordance with the DSM-5 diagnostic criteria, having stabilized medications used for ADHD, being open to communication, and being able to understand and follow instructions at a basic level

Exclusion Criteria:

* having any neurological, orthopedic or psychiatric diagnosis in addition to ADHD diagnosis, having undergone any surgical intervention in the last 3 months, being inadequate in understanding visual and auditory commands, and having a visual or hearing impairment.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Dynamic Occupational Therapy Cognitive Assessment (DOTCA-Ch) | 1 month
  The Dynamic Occupational Therapy Cognitive Assessment (DOTCA-Ch): It was developed to evaluate the cognitive functions of children between the ages of 6 and 12. It includes 22 subtests in 5 cognitive areas; orientation, spatial perception, praxis, visuomotor construction and thinking operations. There is a structured 5-stage scoring system for each subtest. The purpose of the assessment is to identify the child's strengths and deficiencies in different cognitive areas, to measure learning potential and to identify the child's thinking strategies using dynamic procedures. The practice time is approximately 1½ hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No